CLINICAL TRIAL: NCT03906461
Title: LSI (Lesion Index) Workflow Post-Market Observational Study
Brief Title: LSI (Lesion Index) Workflow Observational Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10276
Record Dates: First submitted 2019-03-29; First posted 2019-04-08 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Radiofrequency Ablation — The Tacticath Contact Force Ablation Catheter, Sensor Enabled (TactiCath SE) is designed to facilitate electrophysiological mapping of the heart chambers and to transmit radiofrequency (RF) current to the catheter tip electrode for intracardiac ablation purposes.

SUMMARY:
This clinical study is a prospective, multicenter, post-market, single-arm, observational study designed to characterize the usage of the Lesion Index (LSI) with the market-released TactiCath Contact Force Ablation Catheter, Sensor Enabled (TactiCath SE) in subjects with Paroxysmal Atrial Fibrillation (PAF) in a real-word environment.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize LSI achieved values for durable lesion formation using the TactiCath SE catheter in the different anatomical regions around the pulmonary veins (PVs) of the heart during RF ablation for the treatment of drug-refractory paroxysmal atrial fibrillation (PAF)

Secondary objectives of this study are as follows:

* To characterize the use of EnSite Automap and AutoMark module software settings, including LSI threshold (OUS), contact force, time, power, flow, and AutoMark spacing using the TactiCath SE catheter for RF ablation for the treatment of drug-refractory PAF.
* To characterize LSI achieved values for lesions that reconnected versus those that were durable, both in an acute procedural setting as well as in patients who undergo additional ablations during the 12-month follow-up period after an index RF ablation procedure for the treatment of drug-refractory PAF.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation related procedure.
2. Subject is at least 18 years of age.
3. Subject is willing and able to comply with the protocol-described evaluations and follow-up schedule.
4. Subject plans to undergo a pulmonary vein isolation (PVI) procedure due to symptomatic paroxysmal AF using RF ablation.
5. Subject is refractory or intolerant to at least one class I or class III anti-arrhythmic drug.

   * For the purposes of this study, "intolerant" includes either:

     1. Subject attempted the drug at any dose and either the subject or their physician chose to discontinue for any reason.
     2. Subject was offered the drug and refused to take for any reason.

Exclusion Criteria:

1. Previous ablation or surgery in the left atria.
2. Has an implantable cardiac defibrillator (ICD) (pacemakers without defibrillation capacity are allowable).
3. Participation in another clinical investigation that may confound the results of this study.
4. Pregnant or nursing.
5. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
6. Life expectancy less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll male and female subjects undergoing their first ablation procedure from the documented drug-refractory, paroxysmal atrial fibrillation (PAF) population. Subjects must meet all eligibility criteria and provide written informed consent prior to conducting any investigation-specific procedures not considered standard of care.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Ruffner, PhD, Study Director — EP Program Director
Locations (9):
- United States (4):
  - Mills-Peninsula Medical Center, Burlingame, California
  - St. Vincent Hospital, Indianapolis, Indiana
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Maimonides Medical Center, Brooklyn, New York
- St. Johannes Hospital, Dortmund, Germany
- Ospedale Santa Maria del Prato, Feltre, Italy
- Japan (2):
  - Tokyo Medical and Dental University Hospital of Medicine, Bunkyō-Ku, Tokyo
  - The Jikei University Katsushika Medical Center, Katsushikachō, Tokyo
- Hospital Universitario de Monteprincipe, Boadilla del Monte, Spain

IPD SHARING:
Plan to Share IPD: Undecided
TBD via publication plan

RESULTS

PARTICIPANT FLOW:
Groups:
- TactiCath SE and LSI: Catheter ablation to achieve pulmonary vein isolation using TactiCath SE catheter and the EnSite AutoMark module.
  US only: Operators used their standard metrics for AutoMark. OUS: Operators used LSI as the color metric for AutoMark
Period: Enrollment to Completed Procedure
Arm/Group | TactiCath SE and LSI
Started | 143
Completed | 143
Not Completed | 0
Period: Completed 12-month Follow-up
Arm/Group | TactiCath SE and LSI
Started | 143
Completed | 133
Not Completed | 10
Not completed — Withdrawal by Subject | 4
Not completed — Missed Visit | 6

BASELINE CHARACTERISTICS:
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 91
  More than one race | 1
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 56
  Japan | 30
  Italy | 22
  Germany | 13
  Spain | 22
Hypertension [Count of Participants; unit: Participants] | 83
Pacemaker or implantable cardiac monitor [Count of Participants; unit: Participants] | 2
Procedure to occlude or close left atrial appendage [Count of Participants; unit: Participants] | 0
History of other arrhythmia [Count of Participants; unit: Participants] | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Achieved Lesion Index (LSI) Values
Description: The primary endpoint is a summary of Lesion Index (LSI) values achieved for radiofrequency ablation catheter lesion formation in different anatomical regions of the heart around the pulmonary veins (PVs). LSI is a proprietary index that combines contact force, radiofrequency duration, and radiofrequency current into a single value to express the gradual growth of lesion formation with increasing LSI values.
Time Frame: At time of procedure
Population: LSI achieved values were not available for all subjects. Data may be missing because the LSI algorithm requires six seconds of force and current data as input to report an LSI value or the case files were not received from the site.
Measure: Mean (Standard Deviation); unit: Lesion Index
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 137
Lesion Index
  LSI of Lesions in Anterior Portion of Left Superior Pulmonary Vein | 4.9 (1.0)
  LSI of Lesions in Posterior Portion of Left Superior Pulmonary Vein | 4.8 (1.0)
  LSI of Lesions in Anterior Portion or Left Inferior Pulmonary Vein | 4.9 (1.0)
  LSI of Lesions in Posterior Portion of Left Inferior Pulmonary Vein | 4.7 (1.0)
  LSI of Lesions in Anterior Portion of Right Superior Pulmonary Vein | 5.1 (1.0)
  LSI of Lesions in Posterior Portion of Right Superior Pulmonary Vein | 5.0 (1.0)
  LSI of Lesions in Anterior Portion of Right Inferior Pulmonary Vein | 4.9 (1.1)
  LSI of Lesions in Posterior Portion of Right Inferior Pulmonary Veins | 5.1 (1.0)

2. Secondary Outcome: Ensite AutoMark Settings and Characteristics: Time and AutoMark Time Parameters
Description: Descriptive summary of EnSite AutoMark module software settings and characteristics, including time and AutoMark Time parameters for each lesion. Away time refers to the maximum amount of time the catheter can remain away from the AutoMark region before a new AutoMark will be placed. The AutoMark minimum lesion time refers to the minimum amount of time the catheter tip must remain within the AutoMark region before an AutoMark lesion is placed.
Time Frame: At time of procedure
Population: LSI achieved values were not available for all subjects. Data may be missing because the LSI algorithm requires six seconds of force and current data as input to report an LSI value or the case files were not received from the site. The AutoMark settings and characteristics of all lesions in the subjects with LSI data were analyzed.
Measure: Mean (Standard Deviation); unit: s
Units Other Than Participants: lesions
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 137
Number analyzed (lesions) | 12940
s
  Duration | 14.4 (9.3)
  AutoMark Away Time Parameter | 7.1 (2.2)
  AutoMark Min Lesion Time Parameter | 3.2 (0.9)

3. Secondary Outcome: Ensite AutoMark Settings and Characteristics: Average RF Power Delivered
Description: Descriptive summary of EnSite AutoMark module software settings and characteristics, including average radiofrequency (RF) power delivered for each lesion
Time Frame: At time of procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: W
Units Other Than Participants: lesions
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 137
Number analyzed (lesions) | 12940
W | 38.0 (8.3)

4. Secondary Outcome: Ensite AutoMark Settings and Characteristics: Contact Force
Description: Descriptive summary of EnSite AutoMark module software settings and characteristics, including contact force for each lesion
Time Frame: At time of procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g
Units Other Than Participants: lesions
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 137
Number analyzed (lesions) | 12939
g | 11.7 (7.4)

5. Secondary Outcome: Ensite AutoMark Settings and Characteristics: AutoMark Lesion Spacing Parameter
Description: Descriptive summary of EnSite AutoMark module software settings and characteristics, including AutoMark Lesion Spacing parameter for each lesion
Time Frame: At time of procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: lesions
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 137
Number analyzed (lesions) | 12940
mm | 5.7 (1.7)

6. Secondary Outcome: Number of Participants With Acute Electrical Isolation of Pulmonary Veins
Description: Acute electrical isolation of the pulmonary veins (PVs), 20 minutes after the last RF ablation in the PV region. The number of participants with acute electric isolation of all pulmonary veins is reported.
Time Frame: 20 minutes after last RF ablation in PV region
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants | 143

7. Secondary Outcome: Number of Participants With 7-Day Device or Procedure Related SAEs
Description: Device- or procedure-related SAEs within 7-days of the index procedure
Time Frame: within 7-days of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants | 1

8. Secondary Outcome: Number of Participants With 12-Month Device or Procedure Related SAEs
Description: Device- or procedure-related SAEs within 12-months of index procedure
Time Frame: between 7 days and 12-months of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants | 1

9. Secondary Outcome: Number of Participants With Freedom From AF/AFL/AT Recurrence
Description: Freedom from documented AF/AFL/AT recurrence at 12-months post index ablation, excluding a 90-day blanking period. Freedom from AF/AFL/AT recurrence is defined as no documented episodes greater than 30 seconds with a 24-hour Holter.
Time Frame: No documented episodes greater than 30 seconds with a 24hour-Holter
Population: Analysis population includes subjects with 12 Month visit complete and 24-hour Holter data available.
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 117
Participants | 112

10. Secondary Outcome: Number of Participants With Repeat Ablation
Description: Participants with a repeat ablation up to 12-months post index procedure (excluding 90-day blanking period)
Time Frame: 12-months post index procedure (excluding 90-day blanking period)
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants | 3

11. Secondary Outcome: Number of Participants That Required Touch up Ablation in Each Region
Description: Participants with regions that required touch up ablation.
Time Frame: At time of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants
  Anterior Portion of Left Superior Vein | 5
  Posterior Portion of left Superior Vein | 7
  Posterior Portion of Left Inferior Vein | 5
  Anterior Portion of Left Inferior Vein | 5
  Posterior Portion of Right Superior Vein | 3
  Anterior Portion of Right Superior Vein | 7
  Anterior Portion of Right Inferior Vein | 3
  Posterior Portion of Right Inferior Vein | 3

12. Secondary Outcome: Number of Participants in Which Pulmonary Veins Required Touch-up Ablation
Description: Participants that required touch-up ablation of each pulmonary vein (PV).
Time Frame: At time of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants
  Left Superior Vein | 11
  Left Inferior Vein | 7
  Right Superior Vein | 9
  Right Inferior Vein | 6

13. Secondary Outcome: Number of Participants That Required Index Procedure Touch-up Ablations
Description: Participants who required at least one touch-up ablation during the index procedure
Time Frame: At time of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants | 34

14. Secondary Outcome: LSI Achieved Values for Repeat RF Ablations
Description: In participants who undergo any repeat RF ablation procedures up to 12-months post index procedure, characterization of LSI achieved values for lesions that resulted in electrically conducting gaps versus those that were durable
Time Frame: up to 12-months post index procedure, characterization of LSI achieved values for lesions that resulted in electrically conducting gaps versus those that were durable
Population: The analysis population would include only those subjects with repeat RF ablation procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 3
Participants | NA — There was an insufficient number of participants with events.

15. Secondary Outcome: Overall Procedure Time
Description: Overall procedure time and the subset of time elapsed for: first-pass PVI, any other ablations, and any touch-up ablations
Time Frame: At time of procedure
Population: Analysis population includes all subjects for total initial PV isolation time and total procedure time. Total time for touch-up includes those subjects in which touch-up time was reported. Total non-PV ablation time includes those subjects in which non-PV ablation was done and time was reported.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
minutes
  Total initial PV isolation time | 55.6 (31.2)
  Total time for touch-up: number analyzed (Participants) | 31
  Total time for touch-up | 7.4 (7.8)
  Total non-PV ablation time: number analyzed (Participants) | 52
  Total non-PV ablation time | 22.5 (34.7)
  Total procedure time | 142.5 (53.1)

16. Secondary Outcome: Overall RF Ablation Time
Description: Overall RF ablation time and the subset of RF ablation time for: first-pass PVI, any other ablations, and any touch-up ablations
Time Frame: At time of procedure
Population: Analysis population included all subjects in which RF energy was delivered. Total touch-up RF time only includes subjects in which touch-up ablation was done during the index procedure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
minutes
  Total RF time for initial PVI | 19.3 (9.0)
  Total touch-up RF time: number analyzed (Participants) | 34
  Total touch-up RF time | 2.6 (3.3)
  Total RF time for entire procedure | 22.1 (10.3)

17. Secondary Outcome: Overall Fluoroscopy Time
Description: Overall fluoroscopy time
Time Frame: At time of procedure
Population: Analysis includes subjects in which fluoroscopy was used during the procedure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 127
minutes | 23.7 (20.0)

18. Secondary Outcome: Quality of Life Changes 6-Month
Description: Changes in 5-level EQ-5D (EQ-5D-5L) and AFEQT (Atrial Fibrillation Effect on QualiTy-of-life) quality of life scores at 6-months post index ablation, compared to baseline scores.
  AFEQT scores range from 0 (most severe symptoms) to 100 (no limitation or disability). A positive change indicates an improvement in AF condition.
  EQ-5D-5L EQ VAS scores range from 0 (worst) to 100 (best). A positive change indicates an improvement.
Time Frame: 6 months post index ablation, compared to baseline scores
Population: Analysis population includes those subjects with quality of life scores assessed at both baseline and 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 140
score on a scale
  Change in overall AFEQT Baseline to 6 months | 20.8 (21.9)
  Change in EQ-5D-5L EQ VAS Baseline to 6 months | 6.3 (15.3)

19. Secondary Outcome: Quality of Life Changes 12-Month
Description: Changes in 5-level EQ-5D (EQ-5D-5L) and AFEQT (Atrial Fibrillation Effect on QualiTy-of-life) quality of life scores at 12-months post index ablation, compared to baseline scores.
  AFEQT scores range from 0 (most severe symptoms) to 100 (no limitation or disability). A positive change indicates an improvement in AF condition.
  EQ-5D-5L EQ VAS scores range from 0 (worst) to 100 (best). A positive change indicates an improvement.
Time Frame: 12-months post index ablation, compared to baseline scores
Population: Analysis population includes subjects with Quality of Life scores at both baseline and 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 133
score on a scale
  Change in overall AFEQT score from baseline to 12 months | 23.8 (20.3)
  Change in EQ-5D-5L EQ VAS from Baseline to 12 months | 7.6 (14.2)

20. Secondary Outcome: Number of Participants on Antiarrhythmic Drugs
Description: Antiarrhythmic drug use at 12-months
Time Frame: 12-months
Population: Analysis includes subjects that completed the 12-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 133
Participants | 52

21. Secondary Outcome: Number of Participants With Health Care Utilization
Description: Health care utilization (including number of unscheduled hospital outpatient/ER visits and inpatient hospitalizations due to arrhythmias) collected throughout the 12-month follow-up period
Time Frame: collected throughout the 12-month follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE and LSI
Number analyzed (Participants) | 143
Participants | 13

ADVERSE EVENTS:
Time Frame: 12 months
Description: Per protocol, only device or procedure-related serious adverse events were collected and reported. While defined in the protocol, non-serious and non-related adverse event data was not collected in this study. Determination of whether there was a reasonable possibility that an investigational product or device under investigation caused or contributed to an SAE was determined by the investigator.
Arm/Group | TactiCath SE and LSI
All-Cause Mortality (participants affected / at risk) | 1/143
Serious Adverse Events (participants affected / at risk) | 1/143
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TactiCath SE and LSI (N=143)
Cardiac Perforation or Tamponade (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of study results will be made as a joint multi-center publication with investigators from all sites contributing data. Institutions may publish data and results individually from its site after any of the following (1) a multi-center publication is published, (2) no multicenter publication is submitted within eighteen months after closures of the Study at all sites or (3) sponsor confirms in writing there will be no multi-center publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03906461/Prot_SAP_000.pdf